CLINICAL TRIAL: NCT00159705
Title: A Randomized Placebo-Controlled Trial of the Efficacy and Safety of Pregabalin in the Treatment of Subjects With Neuropathic Pain Associated With Lumbo-Sacral Radiculopathy
Brief Title: Trial of Efficacy and Safety of Pregabalin in Subjects With Neuropathic Pain Associated With Lumbo-Sacral Radiculopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081007
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2008-10

CONDITIONS: Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Pregabalin

INTERVENTIONS:
Drug: pregabalin

SUMMARY:
Trial will evaluate the efficacy and safety of pregabalin in the treatment of subjects with neuropathic pain associated with lumbo-sacral radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Pain consistent with a diagnosis of chronic lumbo-sacral radiculopathy due to spinal stenosis or disk herniation.
* Radicular pain must be present for at least 3 months and pain stable for at least 4 weeks.

Exclusion Criteria:

* Surgery for lumbo-sacral radiculopathy within previous 6 months and/or more than one previous spinal surgery for pain-radiculopathy.
* Epidural injection for lumbo-sacral radiculopathy within previous 6 weeks and/or anticipated need for treatment with opioid analgesics, anti-epileptic medications or tricyclic antidepressants to alleviate pain due to lumbo-sacral radiculopathy during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2005-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Pain measurement

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (12):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Independence, Missouri
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Valley Stream, New York
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
- Belgium (4):
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Eeklo
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Pellenberg
- Canada (7):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Fleurimont, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- Germany (7):
  - Pfizer Investigational Site, Bremen
  - Pfizer Investigational Site, Eichstätt
  - Pfizer Investigational Site, Göppingen
  - Pfizer Investigational Site, Kiel
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Nuremberg
  - Pfizer Investigational Site, Wiesbaden
- Italy (6):
  - Pfizer Investigational Site, Localita' Cravino, Pavia
  - Pfizer Investigational Site, Imperia
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Roma
- Spain (5):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Granada
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Seville
  - Pfizer Investigational Site, Valencia
- Sweden (6):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Lidingö
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Luleå
  - Pfizer Investigational Site, Skellefteå
  - Pfizer Investigational Site, Stockholm
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Inciraltı, İzmir
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081007&StudyName=Trial%20of%20Efficacy%20and%20Safety%20of%20Pregabalin%20in%20Subjects%20with%20Neuropathic%20Pain%20Associated%20with%20Lumbo-Sacral%20Radiculopathy